CLINICAL TRIAL: NCT00710866
Title: Influenza Vaccine Dose-Response in Infants and Toddlers: Immunogenicity and Reactogenicity
Acronym: TITRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Centre for Disease Control (Other Government)
Responsible Party: Dr. Danuta M. Skowronski, BC Centre for Disease Control
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PHAC 6273-15-2008/4160872
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: Influenza Vaccines; Infant; Dose-Response Relationship, Immunologic
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 2 doses 0.5mL VAXIGRIP® at months 0, 1
  Interventions: Biological: Inactivated Influenza Vaccine Trivalent Types A and B (Split Virion)
- 2 (Active Comparator): 2 doses 0.25mL VAXIGRIP® at months 0, 1
  Interventions: Biological: Inactivated Influenza Vaccine Trivalent Types A and B (Split Virion)

INTERVENTIONS:
Biological: Inactivated Influenza Vaccine Trivalent Types A and B (Split Virion) — Arm 1 (experimental group) received two spaced injections of the 0.5 mL (full) dose while arm 2 (comparison group) received the currently recommended two spaced injections of 0.25mL (half) dose of trivalent inactivated split virion influenza vaccine (VAXIGRIP®) manufactured by Sanofi Pasteur, Lyon, France.
  Other Names: VAXIGRIP®

SUMMARY:
The purpose of this study is to compare the antibody response and reaction rates in children age 6-23 months when they are given either the currently recommended schedule of two 0.25ml doses of influenza vaccine one month apart or two 0.5ml doses of influenza vaccine, one month apart.

ELIGIBILITY:
Inclusion Criteria:

* Child healthy (stable chronic conditions acceptable) as established by health assessment interview and verbal history-directed health examination
* Child between and including 6 months of age and 23 months of age (up to and including the day before 24 months of age)
* Child is available and can complete all relevant procedures during the entire study period
* Parent or legal guardian is available and can be reached by phone during the entire study period
* Parent/guardian provides written informed consent
* Parent/guardian is fluent in English

Exclusion Criteria:

* Child has history of laboratory-confirmed influenza
* Child has history of any prior influenza immunization
* Child has history of anaphylactic reaction to any component of the vaccine (i.e. egg)
* Child has received immune globulin or other blood products within the prior six weeks
* Child has received injected or oral steroids within the prior six weeks (inhaled or topical steroids allowed)
* Child has a bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection (thrombocytopenia, coagulation disorder, anti-coagulant therapy)
* Child is or will be enrolled in any other clinical trial of a drug, vaccine or medical device during the study period
* Child is scheduled to receive a live vaccine (notably measles, mumps, rubella or varicella vaccines) during the study period
* Child has a health condition which, in the opinion of the investigator, would interfere with the evaluation or pose a health risk to the child

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 262 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danuta M Skowronski, MD, Principal Investigator — BC Centre for Disease Control
Locations (5):
- Canada (5):
  - Coquitlam, British Columbia
  - Vaccine Evaluation Centre, Vancouver, British Columbia
  - Dalhousie University / IWK Health Centre, Halifax, Nova Scotia
  - McGill University Health Centre - Vaccine Study Centre, Montreal, Quebec
  - Université de Laval - Unité de recherche en santé publique, Québec, Quebec

REFERENCES:
- [Derived] Skowronski DM, Hottes TS, De Serres G, Ward BJ, Janjua NZ, Sabaiduc S, Chan T, Petric M. Influenza Beta/Victoria antigen induces strong recall of Beta/Yamagata but lower Beta/Victoria response in children primed with two doses of Beta/Yamagata. Pediatr Infect Dis J. 2011 Oct;30(10):833-9. doi: 10.1097/INF.0b013e31822db4dc. PMID 21857263
- [Derived] Skowronski DM, Hottes TS, Chong M, De Serres G, Scheifele DW, Ward BJ, Halperin SA, Janjua NZ, Chan T, Sabaiduc S, Petric M. Randomized controlled trial of dose response to influenza vaccine in children aged 6 to 23 months. Pediatrics. 2011 Aug;128(2):e276-89. doi: 10.1542/peds.2010-2777. Epub 2011 Jul 18. PMID 21768314

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5mL VAXIGRIP®: 2 doses 0.5mL VAXIGRIP® at months 0, 1
- 0.25mL VAXIGRIP®: 2 doses 0.25mL VAXIGRIP® at months 0, 1
Period: Overall Study
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Started | 133 | 134
Completed | 124 | 128
Not Completed | 9 | 6
Not completed — Protocol Violation | 5 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Failed to meet eligibility | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP® | Total
Number analyzed (Participants) | 124 | 128 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 124 | 128 | 252
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 1.1 (0.4) | 1.1 (0.4) | 1.1 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 71 | 134
  Male | 61 | 57 | 118
Region of Enrollment [Number; unit: participants]
  Canada | 124 | 128 | 252

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Rate Infants (6-11 Months)-A/Brisbane/59/07(H1N1)
Description: Seroprotection rate: HI titers =>40
Time Frame: 27-46 days after the second dose
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 57 | 63
participants | 41 [9.8 to 15.2] | 34 [8.2 to 12.7]

2. Primary Outcome: Seroprotection Rate Toddlers(12-23 Months)-A/Brisbane/59/07(H1N1)
Description: Seroprotection rate: HI titers =>40
Time Frame: 27-46 days after the second dose
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 60 | 59
participants | 54 | 52

3. Primary Outcome: Seroprotection Rate Infants(6-11 Months)-A/Brisbane/10/07(H3N2)
Description: Seroprotection rate: HI titers =>40
Time Frame: 27-46 days after the second dose
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 57 | 63
participants | 43 | 30

4. Primary Outcome: Seroprotection Rate Toddlers(12-23 Months)-A/Brisbane/10/07(H3N2)
Description: Seroprotection rate: HI titers =>40
Time Frame: 27-46 days after the second dose
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 60 | 59
participants | 55 [10.9 to 15.7] | 52 [7.5 to 11.0]

5. Primary Outcome: Seroprotection Rate Infants (6-11 Months)-B/Florida/4/06(Yamagata)
Time Frame: 27-46 days after the second dose
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 57 | 63
participants | 40 [10.8 to 17.1] | 26 [6.7 to 10.6]

6. Primary Outcome: Seroprotection Rate Toddlers (12-23 Months)-B/Florida/4/06(Yamagata)
Description: Seroprotection rate: HI titers =>40
Time Frame: 27-46 days after the second dose
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 60 | 59
participants | 54 | 55

7. Primary Outcome: Adverse Events: Fever After Either Dose - Infants 6-11 Months
Description: Fever defined as temperature >= 38 C
Time Frame: 3 days after immunization
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 61 | 65
participants | 1 | 7

8. Primary Outcome: Adverse Events: Fever After Either Dose - Toddlers(12-23 Months)-
Description: Fever defined as temperature >= 38 C
Time Frame: 3 days after immunization
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Number analyzed (Participants) | 63 | 61
participants | 6 | 9

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited adverse events were recorded using memory aid after immunization for days 0 to 7 after each injection; reports shown for days 0 to 3 after either injection.
Arm/Group | 0.5mL VAXIGRIP® | 0.25mL VAXIGRIP®
Serious Adverse Events (participants affected / at risk) | 0/124 | 1/128
Other Adverse Events (participants affected / at risk) | 108/124 | 107/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5mL VAXIGRIP® (N=124) | 0.25mL VAXIGRIP® (N=128)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5mL VAXIGRIP® (N=124) | 0.25mL VAXIGRIP® (N=126)
Redness (Skin and subcutaneous tissue disorders) | 28 (28) | 26 (26)
Swelling (Skin and subcutaneous tissue disorders) | 19 (19) | 11 (11)
Induration (Skin and subcutaneous tissue disorders) | 17 (17) | 8 (8)
Tenderness (Skin and subcutaneous tissue disorders) | 28 (28) | 33 (33)
Fever (General disorders) | 11 (11) | 19 (19)
Irritability (General disorders) | 74 (74) | 77 (77)
Decreased appetite (General disorders) | 48 (48) | 55 (55)
Drowsiness (General disorders) | 49 (49) | 53 (53)
Sleep disturbance (General disorders) | 68 (68) | 64 (64)
Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 15 (15)
Ocular (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 8 (8) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Teething (Musculoskeletal and connective tissue disorders) | 13 (13) | 12 (12)
Miscellaneous (General disorders) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No